CLINICAL TRIAL: NCT03819257
Title: Evaluation of Anorectal Function in Perianal Crohn's Disease: a Pilot Study.
Brief Title: Anorectal Function in Perianal Crohn's Disease
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GA18/113514
Record Dates: First submitted 2019-01-18; First posted 2019-01-28 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with perianal Crohn's disease.
  Interventions: Diagnostic Test: Endoanal ultrasound; Diagnostic Test: High-resolution anorectal manometry; Diagnostic Test: Balloon expulsion test

INTERVENTIONS:
Diagnostic Test: Endoanal ultrasound — For the assessment of the internal and external anal sphincter integrity. To evaluate fistulas/perianal abscess and seton placement.
Diagnostic Test: High-resolution anorectal manometry — 1. rest - basal anal pressures at rest over 60 s
  2. squeeze - anal pressure during voluntary effort; long squeeze - anal pressure during sustained voluntary effort
  3. cough - anorectal pressure changes during cough
  4. push - anorectal pressure changes during simulated defecation
  5. rectoanal inhibitory reflex - reflex anal response to rectal distension
  6. rectal sensation - assessment of rectal sensitivity to distension.
Diagnostic Test: Balloon expulsion test — A non-latex balloon will be inserted in the rectum after applying lubricating gel. This balloon is then filled with 50ml of warm water. The patient is ask to sit on a commode and to try to expel the device in privacy, while the time is being recorded. The test ends when the patient expelled the balloon or when 3 minutes are reach.

SUMMARY:
Perianal Crohn's disease is a disabling disease associated with increased morbidity and impaired quality of life. It is associated with pain, discharge, fecal incontinence and sexual and psychological impairment. In refractory cases, a stoma may be necessary. A higher prevalence is seen with increasing Crohn's disease duration and appears to vary according to the disease location. The presence of symptoms associated with anorectal dysfunction, such as fecal incontinence, can sometimes poorly correlate with the presence of anal sphincter abnormalities. Moreover, even in patients without symptoms, the presence of anal sphincter abnormalities may have important implications for the future selection of type of delivery, and might even pose a contra-indication for certain types of anorectal surgeries.

Studies evaluating possible chronic complications of perianal Crohn's disease on anorectal function are lacking. There is a need for a better understanding of the chronic complications of this disease, and the role of high-resolution anorectal manometry in diagnosing these abnormalities during follow-up of these patients. This study will evaluate the chronic repercussions of perianal Crohn's disease in patients with a previous anal fistula and/or abscess that has healed and/or is inactive.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 75 year-old patients
2. CD in clinical remission, defined by a Harvey-Bradshaw index <5
3. Perianal CD history, defined by the presence of a perianal fistula and/or abscess that were treated/heal/inactive
4. Perianal Disease Activity Index (PDAI) of ≤4
5. Asymptomatic or symptomatic patients (anorectal symptoms) will be included, as long they fulfill the other inclusion criteria, like for anorectal symptomatic patients having a PDAI≤4
6. Endoanal ultrasound without an image compatible with new/non-treated abscess or perianal fistula
7. Both previous simple or complex perianal fistula (according to the American College of Gastroenterology) will be considered.

Exclusion Criteria:

1. Women with previous vaginal delivery
2. Ileostomy
3. Previous anorectal surgery as hemorrhoidectomy or lateral sphincterotomy
4. Active rectal disease. No rectal involvement will be defined by no previous rectal involvement ever described or if previous involvement, endoscopy within 18 months showing no current involvement
5. Previous or current anal fissure
6. Anal stricture
7. Current or previous rectovaginal fistula (previous/last pelvic MRI).

A previous seton placement, abscess drainage, fistulotomy and lay open fistula are not an exclusion criteria. Patients with a current seton can only be included if the seton was place more than 24 weeks ago, and the endoanal ultrasound does not show any new/non-treated perianal fistula/abscess.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending hospital with diagnosed perianal Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2020-02-22 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
Resting pressure, squeezing pressure, anorectal pressure changes during cough, anorectal pressure changes during simulated defecation, presence of a rectoanal inhibitory reflex and assessment of rectal sensitivity to distension. | 30 minutes
  Evaluated by high-resolution anorectal manometry.
Anal sphincters integrity. | 5 minutes
  Evaluated by endoanal ultrasound.
Ballon expulsion test duration. | 3 minutes

SECONDARY OUTCOMES:
Presence of symptoms suggesting obstructed defection. | 5 minutes
  Prolonged and unsuccessful straining at stool, self-digitation for defecation, sense of incomplete evacuation or sensation of anorectal obstruction/blockage and a stool frequency of less than three times per week.

OTHER OUTCOMES:
Wexner score (fecal incontinence score). | 5 minutes
  5 items score, including solid, liquid, gas incontinence, wearing pads and lifestyle alterations, scored from 0 (normal) to 4 (more severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Derived] Albuquerque A, Casey J, Fairlamb G, Houghton LA, Selinger C. Evaluation of Anorectal Function in Perianal Crohn's Disease: A Pilot Study. J Clin Med. 2021 Dec 16;10(24):5909. doi: 10.3390/jcm10245909. PMID 34945205